CLINICAL TRIAL: NCT03813628
Title: Evaluation of Patient Satisfaction and Color Difference Between Natural Teeth and Monolithic All-ceramic Crowns Fabricated From Zirconia Reinforced Lithium Silicate Ceramics "Celtra Press" Treated With Different Surface Finishing Protocols.
Brief Title: Evaluation of Patient Satisfaction and Color Difference Between Natural Teeth and Monolithic All-ceramic Crowns Fabricated From Celtra Press Treated With Different Surface Finishing Protocols
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nurhan Sayed Saleh Ahmed, Principal investigator - Fixed prosthodontic department, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-23
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Natural Optical Properties
Keywords: celtra press

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- polished celtra press full coverage crowns (Experimental): a full coverage crown in esthetic area made from celtra press ceramic( zirconia reinforced lithium silicate) and finished by just polishing
  Interventions: Other: polished celtra press full coverage crown
- glazed celtra press full coverage crowns (Experimental): a full coverage crown in esthetic area made from celtra press ceramic( zirconia reinforced lithium silicate) and finished by glazing
  Interventions: Other: glazed celtra press full coverage crowns
- contralateral natural teeth (Active Comparator): the poilshed and glazed all ceramic crowns will be compared by the contralateral natural teeth
  Interventions: Other: contralateral natural teeth

INTERVENTIONS:
Other: polished celtra press full coverage crown — a full coverage crown in esthetic area made from celtra press ceramic( zirconia reinforced lithium silicate) and finished by just polishing
  Other Names: polished all ceramic crown
  Arms: polished celtra press full coverage crowns
Other: glazed celtra press full coverage crowns — a full coverage crown in esthetic area made from celtra press ceramic( zirconia reinforced lithium silicate) and finished by glazing
  Other Names: glazed all ceramic crown
  Arms: glazed celtra press full coverage crowns
Other: contralateral natural teeth — the polished and glazed all ceramic crowns will be compared by the contralateral natural teeth
  Arms: contralateral natural teeth

SUMMARY:
investigating the effect of glazing and polishing on the color difference between natural teeth and all ceramic crowns made from celtra press (zirconia reinforced lithium silicate ceramic).

DETAILED DESCRIPTION:
Two groups of patients will be selected according to special inclusion criteria N=5 in each group total of 10 patients, one of the two groups will receive a glazed zirconia reinforced lithium silicate ''celtra press'' crowns and the other group will receive a polished ones of the same material , after crowns delivery color difference (ΔE) between the natural teeth and the celtra press crown will be measured by a spectrophotometer device (intra oral) and patient satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age range of the patients from 20-45 years old; able to read and sign the informed consent document, illiterate patient will be avoided.
* Patients able physically and psychologically to tolerate conventional restorative procedures.
* Patients with no active periodontal or pulpal diseases, having teeth with good restorations.
* Patients with teeth problems indicated for full coverage restoration ( coronal fracture where partial coverage would lack retention, malposed or malformed teeth).
* Patients with root canal treated teeth requiring full coverage restorations with contralatral tooth not filled or fractured.
* Patients willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth.
* Patients with poor oral hygiene and motivation.
* Pregnant women's to avoid any complication that may occur in dental office due to pregnancy or due to injected anesthetic solution.
* Patients with psychiatric problems or unrealistic expectation
* Deep discoloration of abutment .

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
color match | immediately after crown delivery
  Color match will be measured using "United states pulplic health service " system .
  Scale system :
  * Alpha : Excellent colour match and shade between restoration and adjacent tooth, restoration almost invisible
  * Bravo : Slightly mismatching between the restoration and the adjacent tooth, which is in the normal range of tooth colour, translucence, and/or shade
  * Charlie : Obvious mismatch, beyond the normal range
  * Delta : Gross mismatch/aesthetically displeasing colour, shade, and/or translucence

SECONDARY OUTCOMES:
Color difference | immediately after crown delivery
  The color difference (ΔE) will be measured using spectrophotometer

OTHER OUTCOMES:
patient satisfaction | immediately after crown delivery
  Patient satisfaction using Visual Analogue scale- Binary (Satisfied or not satisfied)

IPD SHARING:
Plan to Share IPD: Undecided